CLINICAL TRIAL: NCT04127682
Title: Antibiotic Prescription for Children With Acute Upper Respiratory Tract Infections in Assiut District: An Exploratory Study.
Brief Title: Antibiotic Prescription for Children With Acute Upper Respiratory Tract Infections in Assiut District
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam T. Amin, Physician, Assiut University
Other Study IDs: AMR_PH01
Record Dates: First submitted 2019-10-13; First posted 2019-10-15 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Antibiotic Side Effect

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: Physicians dealing with cases of pediatrics' acute URIs at PHC units either urban or rural, insurance hospitals or Assiut university hospitals.
  Interventions: Other: Antibiotic KAP questionnaire

INTERVENTIONS:
Other: Antibiotic KAP questionnaire — • Self-administered questionnaire will be used and containing following Physician information (age, sex, place of work, specialty, years of experience, place of work, and post graduate studies and trainings), Practice information (number of days for outpatient's practice/week, average number of patients /day and average percentage of children with ARIs/day), Antibiotic prescription practice (using of guidelines and causes of prescribing antibiotics in acute URIs), Knowledge about antibiotic resistance and attendance of any conference or educational activities concerned with antibiotic use during the last year, Attitude as regard antibiotic prescription.

SUMMARY:
Antibiotics are one of the most commonly prescribed drugs in pediatric care all over the world. Over prescription of antibiotics is a major public health problem and the most important factor in the emergence of antibiotic resistance. It is important to study physicians' antibiotic prescribing behavior to understand its determinant and for further planning of appropriate interventions to optimize antibiotic prescription.

DETAILED DESCRIPTION:
Antibiotics are one of the most commonly prescribed drugs in pediatric care all over the world. Over prescription of antibiotics is a major public health problem and the most important factor in the emergence of antibiotic resistance.

In Egypt, a recent study conducted in El-Minya governorate to investigate antibiotic use in PHC centres and in governmental hospitals, revealed that physician prescriptions of antibiotics for ARIs were extremely high as 82% of pediatric visits for ARIs resulted in an antibiotic prescription. Most of these infections are caused by viruses and do not require antibiotic treatment.

Numerous interventions to improve antibiotic prescribing practices have been reported from various countries with varying results. No single intervention appears to have superior efficacy, but combinations of interventions are typically more effective, and strategies that target health care professionals and/or patients (or parents of young children) have achieved success at reducing antibiotic prescriptions for ARIs.

Despite the emergence of antibiotic resistance and international efforts to reduce antibiotic use, prescription still high and inappropriate. Children are a vulnerable group and inappropriate antibiotic prescription may affect their health and may contribute to development of many diseases as allergies beside emergence of antibiotic resistance. Also, most of acute respiratory infections in children are viral infections and they receive antibiotic for it. So,, it is important to study physicians' antibiotic prescribing behavior to understand its determinant and for further planning of appropriate interventions to optimize antibiotic prescription.

ELIGIBILITY:
Inclusion criteria:

1. Physicians dealing with pediatric cases.
2. GPs, pediatrics, or otolaryngology (ENT) residents.

Exclusion criteria:

1. Physician who didn't work at outpatient clinics.
2. Physicians who are specialized and hold a degree.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians dealing with cases of pediatrics' acute URIs at PHC units either urban or rural, insurance hospitals or Assiut university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Physicians knowledge of antibiotic resistance | 6 months
  By self administered questionnaire
Attitude and practice of physicians as regard antibiotic prescription in pediatric cases of acute upper respiratory tract infections. | 6 months
  By self administered questionnaire

SECONDARY OUTCOMES:
Determinants of physicians' antibiotic prescribing behavior in cases of acute upper respiratory tract infection in children. | 6 months
  By self administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Abd El Aty, Study Director — Public Health Department, Faculty of Medicine, Assiut University; Sabra M Ahmed, Study Director — Public Health Department, Faculty of Medicine, Assiut University; Ghada O El-Sadafi, Study Director — Pediatrics department, Faculty of Medicine, Assiut University; Amira F El-Gazzar, Study Director — Public Health Department, Faculty of Medicine, Assiut University; Mariam T Amin, Principal Investigator — Public Health Department, Faculty of Medicine, Assiut University
Locations (1):
- Faculty of medicine- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Tamma PD, Cosgrove SE. Let the games begin: the race to optimise antibiotic use. Lancet Infect Dis. 2014 Aug;14(8):667-668. doi: 10.1016/S1473-3099(14)70809-6. Epub 2014 Jul 9. No abstract available. PMID 25022437
- [Background] Dooling KL, Kandeel A, Hicks LA, El-Shoubary W, Fawzi K, Kandeel Y, Etman A, Lohiniva AL, Talaat M. Understanding Antibiotic Use in Minya District, Egypt: Physician and Pharmacist Prescribing and the Factors Influencing Their Practices. Antibiotics (Basel). 2014 Jun 20;3(2):233-43. doi: 10.3390/antibiotics3020233. PMID 27025746
- [Background] Meeker D, Linder JA, Fox CR, Friedberg MW, Persell SD, Goldstein NJ, Knight TK, Hay JW, Doctor JN. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. JAMA. 2016 Feb 9;315(6):562-70. doi: 10.1001/jama.2016.0275. PMID 26864410
- [Result] Amin MT, Abd El Aty MA, Ahmed SM, Elsedfy GO, Hassanin ES, El-Gazzar AF. Over prescription of antibiotics in children with acute upper respiratory tract infections: A study on the knowledge, attitude and practices of non-specialized physicians in Egypt. PLoS One. 2022 Nov 3;17(11):e0277308. doi: 10.1371/journal.pone.0277308. eCollection 2022. PMID 36327297